CLINICAL TRIAL: NCT06358144
Title: The Impact of Cannabis Edibles Packaging Descriptors on Consumer Appeal, Harm Perceptions and Willingness to Try: Packaging Imagery Experiment
Brief Title: Cannabis Edibles Packaging Imagery Experiment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB00111438; R01DA053209 (NIH)
Record Dates: First submitted 2024-04-05; First posted 2024-04-10 (Actual); Results first posted 2025-06-08 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-03

CONDITIONS: Cannabis Use
Keywords: Tetrahydrocannabinol (THC); cannabis edibles; Product packaging

STUDY DESIGN:
Intervention Model Description: Participants will complete a 15-minute online survey, where they will be randomized to one of five conditions: four intervention conditions with a different image on the package and one without any imagery.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Flavor Imagery (Experimental): Four edible product packages (gummies, chocolate, mints, cookies) with package imagery in a flavor theme.
  Interventions: Behavioral: Packaging imagery
- Animal Imagery (Experimental): Four edible product packages (gummies, chocolate, mints, cookies) with package imagery in an animal theme.
  Interventions: Behavioral: Packaging imagery
- Nature Imagery (Experimental): Four edible product packages (gummies, chocolate, mints, cookies) with package imagery in a nature theme.
  Interventions: Behavioral: Packaging imagery
- Medical Imagery (Experimental): Four edible product packages (gummies, chocolate, mints, cookies) with package imagery in a medical theme.
  Interventions: Behavioral: Packaging imagery
- No Imagery (Control) (Experimental): Four edible product packages (gummies, chocolate, mints, cookies) without any added packaging imagery.
  Interventions: Behavioral: No Imagery (Control)

INTERVENTIONS:
Behavioral: Packaging imagery — Participants in the four intervention conditions will be shown four cannabis edibles packages that have been altered to contain one of the imagery themes. All participants will see the same four products, and each condition will see the products with the same imagery theme.
  Other Names: four cannabis edibles packages
  Arms: Animal Imagery; Flavor Imagery; Medical Imagery; Nature Imagery
Behavioral: No Imagery (Control) — Participants in the control condition will see the same four product packages, but without any added imagery.
  Other Names: No Imagery
  Arms: No Imagery (Control)

SUMMARY:
The purpose of this study is to assess differences in perceptions of product appeal, harm, and subsequent willingness to try cannabis edibles products with/without packaging imagery.

DETAILED DESCRIPTION:
Cannabis edibles are rapidly leading the legal recreational cannabis market. Cannabis edibles present health harms that are not typical of smoked marijuana, including accidental overconsumption of high levels of Tetrahydrocannabinol (THC) . Product packaging plays an important role in influencing perceptions of a product's appeal and potential harm. This experiment will assign participants to view real cannabis edibles packaging edited with one of four images commonly found on real cannabis edibles products, and ask a series of questions to assess perceptions of product appeal and harm. One group of participants will serve as the control and will see the same cannabis edibles packaging without any imagery.

ELIGIBILITY:
Inclusion Criteria:

* US resident
* Aged 18-65, inclusive
* Up to 13% of participants will be those who identify as Black/African American
* Up to 16% of participants will be those who identify as Hispanic
* Approximately 50% of participants will be past year cannabis users
* Was not a participant on the anteceding experiment, Cannabis Edibles Packaging Descriptors Experiment

Exclusion Criteria:

* Does not currently reside in the United States
* Younger than 18 or older than 65
* Does not provide information regarding history of cannabis use
* Otherwise eligible but demographic and/or user group quotas have been met
* Was a participant on the anteceding experiment, Cannabis Edibles Packaging Descriptors Experiment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1260 (Actual)
Dates: Start 2024-05-23 (Actual); Primary Completion 2024-06-19 (Actual); Study Completion 2024-06-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Beth Reboussin, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from online survey panels.
Pre-assignment Details: Approximately 50% of the participants reported using waterpipe within the past year; the remaining 50% of the sample consisted of not-past-year users and never users.
Period: Overall Study
Arm/Group | No Imagery (Control) | Flavor Imagery | Nature Imagery | Medical Imagery | Animal Imagery
Started | 254 | 244 | 245 | 252 | 265
Completed | 254 | 244 | 245 | 252 | 265
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | No Imagery (Control) | Flavor Imagery | Nature Imagery | Medical Imagery | Animal Imagery | Total
Number analyzed (Participants) | 254 | 244 | 245 | 252 | 265 | 1260
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.7 (13.0) | 41.7 (13.2) | 42.6 (13.5) | 40.9 (13.2) | 42.9 (13.2) | 42.2 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 152 | 136 | 148 | 137 | 135 | 708
  Male | 102 | 108 | 97 | 115 | 130 | 552
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 42 | 49 | 49 | 52 | 43 | 235
  Not Hispanic or Latino | 212 | 195 | 196 | 200 | 222 | 1025
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 3 | 4 | 6 | 1 | 19
  Asian | 4 | 10 | 3 | 6 | 1 | 24
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 1 | 1
  Black or African American | 49 | 46 | 54 | 54 | 60 | 263
  White | 178 | 166 | 156 | 158 | 186 | 844
  More than one race | 9 | 4 | 9 | 9 | 6 | 37
  Unknown or Not Reported | 9 | 15 | 19 | 19 | 10 | 72
Region of Enrollment [Number; unit: participants]
  United States | 254 | 244 | 245 | 252 | 265 | 1260

OUTCOME MEASURES:

1. Primary Outcome: Product Appeal Scoring
Description: One item to assess the appeal of the product. Results will be reported as mean for all products within condition.
  Question: How appealing is this product to you? Response options: (0) Not at all appealing to (10) Very appealing
Time Frame: After exposure to product packaging - up to 1 min
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | No Imagery (Control) | Flavor Imagery | Nature Imagery | Medical Imagery | Animal Imagery
Number analyzed (Participants) | 254 | 244 | 245 | 252 | 265
Score on a scale | 5.54 (0.17) | 6.11 (0.18) | 5.73 (0.18) | 5.70 (0.19) | 5.75 (0.18)

2. Primary Outcome: Package Appeal Scoring
Description: One item to assess appeal of the packaging of the product. Results will be reported as mean for all products within condition.
  Question: How appealing is this packaging to you? Response options: (0) Not at all appealing to (10) Very appealing
Time Frame: After exposure to product packaging - up to 1 min
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | No Imagery (Control) | Flavor Imagery | Nature Imagery | Medical Imagery | Animal Imagery
Number analyzed (Participants) | 254 | 244 | 245 | 252 | 265
Score on a scale | 5.67 (0.17) | 6.50 (0.17) | 6.12 (0.17) | 5.73 (0.19) | 6.05 (0.17)

3. Primary Outcome: Product Harm Perceptions (Absolute) Scoring
Description: After exposure to product packaging; 1 min One item to assess participants' opinions of safety of the product. Results will be reported as the number of each type of response.
  Question: How safe do you think it would be to eat the edible in this package? Response options: (1) Completely unsafe, (2) Somewhat unsafe, (3) Somewhat safe, (4) Completely safe
Time Frame: After exposure to product packaging - up to 1 min
Measure: Count of Units; unit: Number of responses on scale 1-4
Units Other Than Participants: Number of responses on scale 1-4
Arm/Group | No Imagery (Control) | Flavor Imagery | Nature Imagery | Medical Imagery | Animal Imagery
Number analyzed (Participants) | 254 | 244 | 245 | 252 | 265
Number analyzed (Number of responses on scale 1-4) | 1014 | 975 | 979 | 1006 | 1060
Number of responses on scale 1-4
  (1) Completely unsafe | 93 | 62 | 70 | 104 | 101
  (2) Somewhat unsafe | 115 | 99 | 113 | 95 | 100
  (3) Somewhat safe | 464 | 447 | 471 | 440 | 467
  (4) Completely safe | 342 | 367 | 325 | 367 | 392

4. Primary Outcome: Package Harm Perceptions (Absolute) Scoring
Description: One item to assess participants' opinions of product safety based on the packaging. Results will be reported as the number of each type of response.
  Question: How much does this packaging make you think this edible is safe to consume? Response options: (1) Not at all; (2) A little; (3) Somewhat; (4) A lot
Time Frame: After exposure to product packaging - up to 1 min
Measure: Count of Units; unit: Number of responses on scale 1-4
Units Other Than Participants: Number of responses on scale 1-4
Arm/Group | No Imagery (Control) | Flavor Imagery | Nature Imagery | Medical Imagery | Animal Imagery
Number analyzed (Participants) | 254 | 244 | 245 | 252 | 265
Number analyzed (Number of responses on scale 1-4) | 1014 | 974 | 1079 | 1007 | 1057
Number of responses on scale 1-4
  (1) Not at all | 162 | 110 | 129 | 126 | 158
  (2) A little | 183 | 152 | 199 | 162 | 157
  (3) Somewhat | 393 | 396 | 467 | 409 | 420
  (4) A lot | 276 | 316 | 284 | 310 | 322

5. Primary Outcome: Willingness to Try Free Sample Scoring
Description: One question will assess the participant's willingness to try the product shown. Results will be reported as the number of each type of response.
  Question: How interested would you be in a free sample of this product? Response options: (1) Not at all; (2) Slightly; (3) Somewhat; (4) Moderately; (5) Very
Time Frame: After exposure to product packaging - up to 1 min
Measure: Count of Units; unit: Number of responses on scale 1-5
Units Other Than Participants: Number of responses on scale 1-5
Arm/Group | No Imagery (Control) | Flavor Imagery | Nature Imagery | Medical Imagery | Animal Imagery
Number analyzed (Participants) | 254 | 244 | 245 | 252 | 265
Number analyzed (Number of responses on scale 1-5) | 1016 | 974 | 980 | 1008 | 1059
Number of responses on scale 1-5
  (1) Not at all | 213 | 205 | 232 | 191 | 238
  (2) Slightly | 105 | 87 | 78 | 71 | 83
  (3) Somewhat | 146 | 148 | 156 | 174 | 146
  (4) Moderately | 184 | 168 | 170 | 176 | 184
  (5) Very | 368 | 366 | 344 | 396 | 408

6. Primary Outcome: Willingness to Try Product Scoring
Description: One item to assess the participants' willingness to try the product based on the packaging. Results will be reported as the number of each type of response.
  Question: How much does seeing this packaging make you want to try this edible? Response options: (1) Not at all; (2) A little; (3) Somewhat; (4) A lot
Time Frame: After exposure to product packaging - up to 1 min
Measure: Count of Units; unit: Number of responses on scale 1-4
Units Other Than Participants: Number of responses on scale 1-4
Arm/Group | No Imagery (Control) | Flavor Imagery | Nature Imagery | Medical Imagery | Animal Imagery
Number analyzed (Participants) | 254 | 244 | 245 | 252 | 265
Number analyzed (Number of responses on scale 1-4) | 1015 | 975 | 977 | 1003 | 1060
Number of responses on scale 1-4
  (1) Not at all | 241 | 201 | 238 | 216 | 272
  (2) A little | 197 | 173 | 176 | 143 | 158
  (3) Somewhat | 295 | 286 | 275 | 329 | 302
  (4) A lot | 282 | 315 | 288 | 315 | 328

7. Secondary Outcome: Appeal to Children Scoring
Description: One item to assess the participants' assessment of the product packaging's potential appeal to children. Results will be reported as mean for all products within condition.
  Question: How appealing do you think this packaging would be to children? Response options: (0) Not at all appealing to (10) Very appealing
Time Frame: After exposure to product packaging - up to 1 min
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | No Imagery (Control) | Flavor Imagery | Nature Imagery | Medical Imagery | Animal Imagery
Number analyzed (Participants) | 254 | 244 | 245 | 252 | 265
Score on a scale | 4.73 (0.17) | 5.62 (0.16) | 4.94 (0.17) | 4.62 (0.17) | 5.87 (0.17)

8. Secondary Outcome: Harm Perceptions (Relative) Scoring
Description: One question assessing participants' opinions of safety of the product compared to other, similar, products. Results will be reported as the number of each type of response.
  Question: Compared to other edible products on the market, how safe do you think the edible in this package is? Response options: (1) Much less safe; (2) Somewhat less safe; (3) As safe; (4) Somewhat safer; (5) Much safer
Time Frame: After exposure to product packaging - up to 1 min
Measure: Count of Units; unit: Number of responses on scale 1-5
Units Other Than Participants: Number of responses on scale 1-5
Arm/Group | No Imagery (Control) | Flavor Imagery | Nature Imagery | Medical Imagery | Animal Imagery
Number analyzed (Participants) | 254 | 244 | 245 | 252 | 265
Number analyzed (Number of responses on scale 1-5) | 1016 | 976 | 979 | 1008 | 1057
Number of responses on scale 1-5
  (1) Much less safe | 79 | 53 | 56 | 84 | 86
  (2) Somewhat less safe | 72 | 54 | 71 | 64 | 62
  (3) As safe | 522 | 469 | 492 | 433 | 526
  (4) Somewhat safer | 210 | 244 | 201 | 226 | 211
  (5) Much safer | 133 | 156 | 159 | 201 | 172

9. Other Pre Specified Outcome: Perception of Quality Scoring
Description: One item to assess the participants' perceptions of the quality of the product. Results will be reported as the number of each type of response.
  Question: To what extent do you agree or disagree that this looks like a good quality product? Response options: (1) Strongly disagree to (5) Strongly agree
Time Frame: After exposure to product packaging - up to 1 min
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Perception of Good Taste Scoring
Description: One item to assess the participants' perceptions of the taste of the product. Results will be reported as the number of each type of response.
  Question: To what extent do you agree or disagree that this edible might taste good? Response options: (1) Strongly disagree to (5) Strongly agree
Time Frame: After exposure to product packaging - up to 1 min
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Perception of Healthfulness of Product Scoring
Description: One item to asses the participants' perceptions of the healthfulness of the product based on the packaging. Results will be reported as the number of each type of response.
  Question: How much does this packaging make you think this edible is healthy? Response options: (1) Not at all; (2) A little; (3) Somewhat; (4) A lot
Time Frame: After exposure to product packaging - up to 1 min
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From the time of consent up to completion of the survey (approximately 1 hour).
Arm/Group | No Imagery (Control) | Flavor Imagery | Nature Imagery | Medical Imagery | Animal Imagery
All-Cause Mortality (participants affected / at risk) | 0/254 | 0/244 | 0/245 | 0/252 | 0/265
Serious Adverse Events (participants affected / at risk) | 0/254 | 0/244 | 0/245 | 0/252 | 0/265
Other Adverse Events (participants affected / at risk) | 0/254 | 0/244 | 0/245 | 0/252 | 0/265

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-02-19): https://cdn.clinicaltrials.gov/large-docs/44/NCT06358144/Prot_SAP_001.pdf
  • Informed Consent Form (2024-04-02): https://cdn.clinicaltrials.gov/large-docs/44/NCT06358144/ICF_000.pdf